CLINICAL TRIAL: NCT00066313
Title: A Phase II Study Of ZD6474 Or Placebo In Small Cell Lung Cancer Patients Who Have Complete Or Partial Response To Induction Chemotherapy +/- Radiation Therapy
Brief Title: ZD6474 in Treating Patients With Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: D4200C00005; CAN-NCIC-BR20; ZENECA-6474IL/0005; CDR0000315518 (Other: Ct.gov temporary)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer; limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — vandetanib; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: vandetanib
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: ZD6474 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. ZD6474 may also stop the growth of small cell lung cancer by blocking blood flow to the tumor.

PURPOSE: This randomized phase II trial is studying how well ZD6474 works compared to placebo in treating patients with small cell lung cancer that has responded to previous chemotherapy with or without radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the progression-free survival of patients with previously treated small cell lung cancer (SCLC) treated with ZD6474 vs placebo.
* Compare the response rate of patients treated with these regimens (only patients who had measurable disease outside a prior radiation field at study entry).
* Compare the toxicity and tolerability of these regimens in these patients.
* Compare the pharmacokinetics of these regimens in these patients.
* Correlate outcome and response with vascular endothelial growth factor expression and microvessel density in patients treated with these regimens.
* Compare the quality of life of patients treated with these regimens.
* Provide a comprehensive tumor, plasma, and urine bank linked to a clinical database for further study of molecular markers in SCLC.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to participating center, timing of prior radiotherapy (early [before day 1, course 4 of chemotherapy] vs late vs no prior radiotherapy), stage of disease at diagnosis (limited vs extensive), and response at study entry (complete vs partial). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral ZD6474 daily.
* Arm II: Patients receive oral placebo daily. In both arms, courses repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, every 4 weeks while on therapy, and then every 8 weeks until disease progression.

Patients are followed every 8 weeks until disease progression and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 100 patients (50 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed small cell carcinoma of the lung

  * Small cell and variant histology allowed
  * No mixed tumors (small and large cell)
  * No neuroendocrine tumors of the lung
* Must have received at least 4 courses of first-line combination chemotherapy as part of an induction regimen

  * No prior change in regimen due to disease progression
* Must have achieved a radiologically confirmed (i.e., CT scan, chest x-ray, or bone scan) complete response (CR) or partial response (PR) after prior chemotherapy with or without radiotherapy AND meets 1 of the following criteria:

  * No more than 28 days since prior chemotherapy
  * At least 7 and no more than 14 days since prior radiotherapy if administered after completion of prior chemotherapy*
* No CNS metastases

  * Asymptomatic patients with CNS metastases who received prior therapeutic cranial irradiation and are on stable, decreasing, or no steroids are eligible
  * No symptomatic lesions or evidence of necrosis or bleeding NOTE: *Randomization may take place up to 21 days after prior radiotherapy in the instance of severe esophagitis that precludes administration of oral medications

PATIENT CHARACTERISTICS:

Age

* Over 16

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No history of bleeding diathesis

Hepatic

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* ALT less than 2.5 times ULN

Renal

* Creatinine less than 1.5 times ULN
* Calcium normal

Cardiovascular

* No prior ventricular arrhythmia that was symptomatic or required treatment (CTC grade 3), including any of the following:

  * Multifocal premature ventricular contractions
  * Bigeminy
  * Trigeminy
  * Ventricular tachycardia
* No prior QT prolongation with any medication
* No congenital long QT syndrome
* No QT and QTc (with Bazett's correction) that is unmeasurable or is 460 msec or higher on screening ECG
* No significant cardiac event, including symptomatic heart failure or angina, within the past 3 months or any cardiac disease that increases the risk for ventricular arrhythmia
* No ongoing chronic atrial fibrillation
* LVEF at least 45% by MUGA for patients with significant cardiac history (myocardial infarction, severe hypertension, or arrhythmia) OR who received prior doxorubicin greater than 450 mg/m^2

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Potassium normal
* Magnesium normal
* No serious active infection
* No recent major bleeding
* No other concurrent serious underlying medical condition that would preclude study participation
* Willing and able to complete quality of life questionnaires in English or French

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior signal transduction inhibitors
* No prior angiogenesis inhibitors
* No concurrent anticancer biologic therapy or immunotherapy

Chemotherapy

* See Disease Characteristics
* Recovered from prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* Recovered from prior radiotherapy
* No concurrent anticancer radiotherapy

  * Concurrent low-dose, nonmyelosuppressive palliative radiotherapy allowed

Surgery

* More than 2 weeks since prior major surgery

Other

* More than 4 weeks since prior investigational drugs
* No prior epidermal growth factor receptor inhibitors
* No prior vascular endothelial growth factor receptor inhibitors
* No concurrent CYP3A4 inhibitors or inducers, including any of the following:

  * Verapamil
  * Rifampin
  * Phenytoin
  * Carbamazepine
  * Barbiturates
  * Hypericum perforatum (St. John's wort)
* No concurrent medication that affects QT/QTc and/or induces torsades de pointes
* No other concurrent anticancer cytotoxic therapy
* No other concurrent investigational drugs during and for 30 days after study participation
* No concurrent oral bisphosphonates (e.g., clodronate)

  * Concurrent IV bisphosphonates allowed
* No concurrent 5HT_3 antagonists

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-05; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Overall Survival
Response rates
Toxicity and safety
Pharmacokinetics
Quality of life (QOL) as measured by EORTC QLQ-C30 and QLQ-LC13

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (21):
- Canada (21):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - Fraser/Valley Cancer Centre at British Columbia Cancer Agency, Surrey, British Columbia
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - Moncton Hospital, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - St. Catharines General Hospital at Niagara Health System, St. Catharines, Ontario
  - Northwestern Ontario Regional Cancer Care at Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Toronto Sunnybrook Regional Cancer Centre at Sunnybrook and Women's College Health Sciences Centre, Toronto, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Windsor Regional Cancer Centre at Windsor Regional Hospital, Windsor, Ontario
  - Hopital Notre- Dame du CHUM, Montreal, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec
  - L'Hopital Laval, Ste-Foy, Quebec
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Arnold AM, Seymour L, Smylie M, Ding K, Ung Y, Findlay B, Lee CW, Djurfeldt M, Whitehead M, Ellis P, Goss G, Chan A, Meharchand J, Alam Y, Gregg R, Butts C, Langmuir P, Shepherd F; National Cancer Institute of Canada Clinical Trials Group Study BR.20. Phase II study of vandetanib or placebo in small-cell lung cancer patients after complete or partial response to induction chemotherapy with or without radiation therapy: National Cancer Institute of Canada Clinical Trials Group Study BR.20. J Clin Oncol. 2007 Sep 20;25(27):4278-84. doi: 10.1200/JCO.2007.12.3083. PMID 17878480